CLINICAL TRIAL: NCT01592708
Title: A Prospective Evaluation of an Anesthesia Protocol to Reduce Post-operative and Post-discharge Nausea and Vomiting in a High Risk Orthognathic Surgery Population
Brief Title: Study of Anesthesia Techniques to Reduce Nausea and Vomiting After Jaw Corrective Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-0622; R01DE005215 (NIH)
Record Dates: First submitted 2012-04-16; First posted 2012-05-07 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-06

CONDITIONS: Post-operative Nausea; Post-operative Vomiting; Nausea Persistent
Keywords: orthognathic surgery; maxillary osteotomy; post operative nausea vomiting; post discharge nausea vomiting; anesthesia
MeSH Terms: interventions — Transdermal Patch; Methylprednisolone Hemisuccinate; Droperidol; Ondansetron; Ketorolac; Ibuprofen; Fentanyl; Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antiemetic anesthesia protocol (Active Comparator): Scopolamine 1.5 milligram(mg) patch Propofol infusion remifentanil infusion 250mg erythromycin po for 2 doses Solumedrol 0.625mg IV droperidol 4mg IV Ondansetron Ketorolac 30mg IV ibuprofen 600mg po q6h Fentanyl Hydrocodone/Tylenol po
  Interventions: Other: Antiemetic anesthesia protocol

INTERVENTIONS:
Other: Antiemetic anesthesia protocol — Intervention group consisted of patients undergoing maxillary osteotomy who received an antiemetic protocol designed to provide multimodal antiemetic therapy which have been shown to help prevent and/or treat postoperative nausea, combined with the elimination of anesthetic factors that may contribute to postoperative nausea and vomiting.
  Other Names: Scopolamine 1.5 milligram(mg) patch; Propofol infusion; remifentanil infusion; 250mg erythromycin po for 2 doses; Solumedrol; 0.625mg IV droperidol; 4mg IV Ondansetron; Ketorolac 30mg IV; ibuprofen 600mg po q6h; Fentanyl; Hydrocodone/Tylenol po

SUMMARY:
The purpose of this study is to determine whether a multi-modal anesthesia and pain control protocol reduces post-operative and post-discharge nausea and vomiting (PONV and PDNV) in patients undergoing upper jaw corrective surgery.

DETAILED DESCRIPTION:
Post-operative and post-discharge nausea and vomiting (PONV and PDNV) plague post-anesthesia and surgical care. This fact remains especially true for the orthognathic surgery (OS) population undergoing procedures involving the maxilla. Current data estimate that the incidence of PONV for OS patients undergoing surgery involving the maxilla is between 44% and 68% as compared to 8% to 30% in general surgical populations, despite application of conventional therapies. No one has accounted for or addressed this difference in clinical outcomes.

The implications of PONV for both individual health and overall health care system function are considerable. For individual patients, PONV can result in dehydration, wound dehiscence, intra-oral bleeding with continued swallowing of blood, significant anxiety and agitation (particularly for OS patients who often have heavy elastics closing their jaws together after surgery), and, in extreme cases, esophageal damage or the risk of pulmonary aspiration. Evidence shows fear of PONV overshadows concerns about pain in surgical patients. At the health care system level, evidence suggests PONV can significantly increase health care costs through prolonged post-anesthesia care unit (PACU) stays and unplanned hospital admissions following outpatient procedures. In one seminal study the odds ratio for unplanned admission due to vomiting after intended outpatient surgery was 3.4, an alarmingly high figure exceeded only by the odds ratios for readmission due to pain or bleeding.

Established patient-related risk factors for PONV include female gender, tobacco abstinence, and history of prior PONV or motion sickness; additional patient factors may include younger age, low American Society of Anesthesiologists Physical Status Classification System status, anxiety, and a migraine headache history. Known anesthesia technique-related risk factors include volatile anesthetic and nitrous oxide use as well as excessive IV opioid administration. High dose neuromuscular blockade reversal agents have also been implicated. Surgery-related factors include duration of surgery and type of surgery, with OS ranking among the high-risk types.

Because PONV (and PDNV) prevention and treatment for the OS population remain under-investigated domains of clinical care, the investigators seek to address this deficiency through multi-modal prophylactic therapy. As more OS procedures are performed, many on an ambulatory basis, tactics to reduce the high incidence of PONV in this surgical population become important to maximize patient safety and satisfaction and to contain costs.

The investigators' protocol will synthesize several recommendations to reduce risk of PONV. Volatile anesthetics and nitrous oxide will be avoided in favor of a total intravenous (IV) anesthetic involving propofol, neostigmine will be minimized, hydration goals will be set, and opioid sparing analgesics will be utilized. It is recommended that patients at high risk for PONV receive combination therapy with prophylactic agents from multiple classes. Among those shown to reduce PONV are 5-HT3 receptor antagonists (such as ondansetron), droperidol, and dexamethasone. Transdermal (TD) scopolamine is another effective adjunctive therapy to reduce PONV. Additionally, the investigators posit that the constant swallowing of small amounts of oozing blood and its retention in the stomach following OS contribute to the high incidence of PONV and PDNV in the OS population. Thus sub-bacteriostatic doses of erythromycin, capitalizing on erythromycin's established properties as a motilin agonist and thus a pro-kinetic, will be added to the evidence-based multi-modal regimen. Erythromycin has been chosen over metoclopramide due to safety profile and its well-characterized impact on gastric motility and even PONV.

Rescue anti-nausea and anti-emetic therapy will be chosen from several options at the discretion of the treating physician. Options that work through several mechanisms have been selected based on the Society of Ambulatory Anesthesia Guidelines and on data from a randomized, double-blind, placebo-controlled study of over 2000 subjects.

Anesthesia variables as well as post-operative analgesic regimens are the primary targets of the investigators' multimodal regimen. Multimodal therapy has been shown to be superior to single agent therapy. One particularly compelling example showed a 98% response rate (no PONV) vs 76% among those receiving mono-therapy and 59% receiving routine anesthesia with placebo. Despite these reported successes, PONV remains a major problem for patients undergoing OS and many other procedures. This study represents one step towards understanding and addressing this significant peri-operative problem.

This proposed study will compare a cohort receiving a multimodal regimen with a retrospective control cohort reviewed in an IRB-approved study at the same institution. The investigators' re-use of the data adds no risk of harm or disclosure to the control subjects. Utilization of this retrospective control has an important advantage over a concurrent control: It allows comparison to a group treated at the same institution without the potential introduction of bias by alerting practitioners to the extent of the PONV problem in OS. The investigators believe that, as the under-recognition of the OS group as high-risk likely contributes to the high rate of PONV these patients experience, education of the anesthesia community introduces a potential confounding variable. Further, comparing practice "as is" to the proposed protocol maximizes generalizability to other institutions. If, as anticipated, significant reductions in PONV and PDNV experience are found, prospective randomized trials to tease out nuances of contributing factors could be undertaken.

Potential influencing patient- and surgery-related variables will be collected to allow comparison of the two cohorts using logistic regression analyses.

Even less well understood than PONV is PDNV; additional studies are needed to deepen understanding of the risk factors and treatment options for PDNV. A prior study from the investigators' institution demonstrated a high incidence of PDNV in the OS population - 43% experienced nausea and 23% vomited after discharge in contrast to general reported rates of 17% PDN and 8% PDV. This study should offer additional insight into PONV's less understood counterpart through diary review of patient's self-reported experience of PDNV following discharge from direct medical supervision.

ELIGIBILITY:
Inclusion Criteria:

* 15 years old or older
* Undergoing elective orthognathic surgery involving a maxillary osteotomy

Exclusion Criteria:

* uncontrolled GERD or hiatal hernia
* glaucoma
* seizure disorder
* COPD
* obstructive sleep apnea
* chronic kidney disease stage III or greater
* known prolonged QT interval (QTc > 460) or the same found incidentally
* history of severe constipation
* pre-existing chronic nausea or vomiting
* allergies or contraindications to protocol medications
* patient insistence on inhalational induction of anesthesia.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ceib Philllips, PhD, MPH, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Silva AC, O'Ryan F, Poor DB. Postoperative nausea and vomiting (PONV) after orthognathic surgery: a retrospective study and literature review. J Oral Maxillofac Surg. 2006 Sep;64(9):1385-97. doi: 10.1016/j.joms.2006.05.024. PMID 16916674
- [Background] Cohen MM, Duncan PG, DeBoer DP, Tweed WA. The postoperative interview: assessing risk factors for nausea and vomiting. Anesth Analg. 1994 Jan;78(1):7-16. doi: 10.1213/00000539-199401000-00004. PMID 8267183
- [Background] Chung F, Un V, Su J. Postoperative symptoms 24 hours after ambulatory anaesthesia. Can J Anaesth. 1996 Nov;43(11):1121-7. doi: 10.1007/BF03011838. PMID 8922767
- [Background] Peacock JE, Philip BK. Ambulatory anesthesia experience with remifentanil. Anesth Analg. 1999 Oct;89(4 Suppl):22. doi: 10.1097/00000539-199910001-00005. No abstract available. PMID 10511074
- [Background] Philip BK. Patients' assessment of ambulatory anesthesia and surgery. J Clin Anesth. 1992 Sep-Oct;4(5):355-8. doi: 10.1016/0952-8180(92)90155-t. PMID 1389187
- [Background] Gan TJ, Meyer T, Apfel CC, Chung F, Davis PJ, Eubanks S, Kovac A, Philip BK, Sessler DI, Temo J, Tramer MR, Watcha M; Department of Anesthesiology, Duke University Medical Center. Consensus guidelines for managing postoperative nausea and vomiting. Anesth Analg. 2003 Jul;97(1):62-71, table of contents. doi: 10.1213/01.ane.0000068580.00245.95. PMID 12818945
- [Background] Watcha MF, White PF. Postoperative nausea and vomiting. Its etiology, treatment, and prevention. Anesthesiology. 1992 Jul;77(1):162-84. doi: 10.1097/00000542-199207000-00023. PMID 1609990
- [Background] Watcha MF, White PF. Post-operative nausea and vomiting: do they matter? Eur J Anaesthesiol Suppl. 1995 May;10:18-23. PMID 7641638
- [Background] Gold BS, Kitz DS, Lecky JH, Neuhaus JM. Unanticipated admission to the hospital following ambulatory surgery. JAMA. 1989 Dec 1;262(21):3008-10. PMID 2810644
- [Background] Koivuranta M, Laara E, Snare L, Alahuhta S. A survey of postoperative nausea and vomiting. Anaesthesia. 1997 May;52(5):443-9. doi: 10.1111/j.1365-2044.1997.117-az0113.x. PMID 9165963
- [Background] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299
- [Background] Gan T, Sloan F, Dear Gde L, El-Moalem HE, Lubarsky DA. How much are patients willing to pay to avoid postoperative nausea and vomiting? Anesth Analg. 2001 Feb;92(2):393-400. doi: 10.1097/00000539-200102000-00022. PMID 11159239
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Fero KE, Jalota L, Hornuss C, Apfel CC. Pharmacologic management of postoperative nausea and vomiting. Expert Opin Pharmacother. 2011 Oct;12(15):2283-96. doi: 10.1517/14656566.2011.598856. Epub 2011 Jul 15. PMID 21756206
- [Background] Gan TJ, Meyer TA, Apfel CC, Chung F, Davis PJ, Habib AS, Hooper VD, Kovac AL, Kranke P, Myles P, Philip BK, Samsa G, Sessler DI, Temo J, Tramer MR, Vander Kolk C, Watcha M; Society for Ambulatory Anesthesia. Society for Ambulatory Anesthesia guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2007 Dec;105(6):1615-28, table of contents. doi: 10.1213/01.ane.0000295230.55439.f4. PMID 18042859
- [Background] Apfel CC, Korttila K, Abdalla M, Kerger H, Turan A, Vedder I, Zernak C, Danner K, Jokela R, Pocock SJ, Trenkler S, Kredel M, Biedler A, Sessler DI, Roewer N; IMPACT Investigators. A factorial trial of six interventions for the prevention of postoperative nausea and vomiting. N Engl J Med. 2004 Jun 10;350(24):2441-51. doi: 10.1056/NEJMoa032196. PMID 15190136
- [Background] Tramer MR, Fuchs-Buder T. Omitting antagonism of neuromuscular block: effect on postoperative nausea and vomiting and risk of residual paralysis. A systematic review. Br J Anaesth. 1999 Mar;82(3):379-86. doi: 10.1093/bja/82.3.379. PMID 10434820
- [Background] Fortney JT, Gan TJ, Graczyk S, Wetchler B, Melson T, Khalil S, McKenzie R, Parrillo S, Glass PS, Moote C, Wermeling D, Parasuraman TV, Duncan B, Creed MR. A comparison of the efficacy, safety, and patient satisfaction of ondansetron versus droperidol as antiemetics for elective outpatient surgical procedures. S3A-409 and S3A-410 Study Groups. Anesth Analg. 1998 Apr;86(4):731-8. doi: 10.1097/00000539-199804000-00011. PMID 9539593
- [Background] Kranke P, Morin AM, Roewer N, Wulf H, Eberhart LH. The efficacy and safety of transdermal scopolamine for the prevention of postoperative nausea and vomiting: a quantitative systematic review. Anesth Analg. 2002 Jul;95(1):133-43, table of contents. doi: 10.1097/00000539-200207000-00024. PMID 12088957
- [Background] Apfel CC, Zhang K, George E, Shi S, Jalota L, Hornuss C, Fero KE, Heidrich F, Pergolizzi JV, Cakmakkaya OS, Kranke P. Transdermal scopolamine for the prevention of postoperative nausea and vomiting: a systematic review and meta-analysis. Clin Ther. 2010 Nov;32(12):1987-2002. doi: 10.1016/j.clinthera.2010.11.014. PMID 21118734
- [Background] Itoh Z, Nakaya M, Suzuki T, Arai H, Wakabayashi K. Erythromycin mimics exogenous motilin in gastrointestinal contractile activity in the dog. Am J Physiol. 1984 Dec;247(6 Pt 1):G688-94. doi: 10.1152/ajpgi.1984.247.6.G688. PMID 6507625
- [Background] Kopp VJ, Mayer DC, Shaheen NJ. Intravenous erythromycin promotes gastric emptying prior to emergency anesthesia. Anesthesiology. 1997 Sep;87(3):703-5. doi: 10.1097/00000542-199709000-00037. No abstract available. PMID 9316982
- [Background] Barkun AN, Bardou M, Kuipers EJ, Sung J, Hunt RH, Martel M, Sinclair P; International Consensus Upper Gastrointestinal Bleeding Conference Group. International consensus recommendations on the management of patients with nonvariceal upper gastrointestinal bleeding. Ann Intern Med. 2010 Jan 19;152(2):101-13. doi: 10.7326/0003-4819-152-2-201001190-00009. PMID 20083829
- [Background] Barkun AN, Bardou M, Martel M, Gralnek IM, Sung JJ. Prokinetics in acute upper GI bleeding: a meta-analysis. Gastrointest Endosc. 2010 Dec;72(6):1138-45. doi: 10.1016/j.gie.2010.08.011. PMID 20970794
- [Background] Habib AS, Gan TJ. The effectiveness of rescue antiemetics after failure of prophylaxis with ondansetron or droperidol: a preliminary report. J Clin Anesth. 2005 Feb;17(1):62-5. doi: 10.1016/j.jclinane.2004.04.004. PMID 15721732
- [Background] Scuderi PE, James RL, Harris L, Mims GR 3rd. Multimodal antiemetic management prevents early postoperative vomiting after outpatient laparoscopy. Anesth Analg. 2000 Dec;91(6):1408-14. doi: 10.1097/00000539-200012000-00020. PMID 11093990
- [Background] Phillips C, Blakey G 3rd. Short-term recovery after orthognathic surgery: a medical daily diary approach. Int J Oral Maxillofac Surg. 2008 Oct;37(10):892-6. doi: 10.1016/j.ijom.2008.07.005. Epub 2008 Sep 2. PMID 18768296
- [Background] Lu CW, Jean WH, Wu CC, Shieh JS, Lin TY. Antiemetic efficacy of metoclopramide and diphenhydramine added to patient-controlled morphine analgesia: a randomised controlled trial. Eur J Anaesthesiol. 2010 Dec;27(12):1052-7. doi: 10.1097/EJA.0b013e32833f53b8. PMID 20829700
- [Background] Kovac AL. Prevention and treatment of postoperative nausea and vomiting. Drugs. 2000 Feb;59(2):213-43. doi: 10.2165/00003495-200059020-00005. PMID 10730546

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Cohort: Patients undergoing maxillary surgery using antiemetic anesthesia protocol
- Comparison Cohort: This arm was a retrospective comparison cohort treated at the same institution, managed per provider preference prior to protocol implementation.
Period: Overall Study
Arm/Group | Intervention Cohort | Comparison Cohort
Started | 96 | 137
Completed | 93 | 137
Not Completed | 3 | 0
Not completed — Protocol Violation | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Cohort: This arm was managed perioperatively with the protocol.
- Total: Total of all reporting groups
Arm/Group | Intervention Cohort | Comparison Cohort | Total
Number analyzed (Participants) | 93 | 137 | 230
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 20 [17 to 24] | 19 [17 to 23] | 19 [17 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 89 | 143
  Male | 39 | 48 | 87

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Nausea
Description: End of surgery time determined by anesthesia portion of the medical record. PONV to be assessed by review of surgeons' and nurses' notes in the medical record as well as through review of patient diaries. Vomiting constitutes a safety issue and, as such, associated adverse events will be noted.
Time Frame: End of surgery to discharge from hospital
Measure: Number; unit: percentage of subjects with PON
Groups:
- Intervention Cohort: Patients undergoing maxillary surgery using the antiemetic anesthetic protocol
Arm/Group | Intervention Cohort | Comparison Cohort
Number analyzed (Participants) | 93 | 137
percentage of subjects with PON | 24 | 70

2. Secondary Outcome: Hospital Length of Stay
Description: Anesthesia start time determined from anesthesia portion of the medical record. Time at which discharge order was placed will serve as time of discharge.
Time Frame: Anesthesia start time to placement of hospital discharge order - average 26 - 28 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Intervention Cohort | Comparison Cohort
Number analyzed (Participants) | 93 | 137
hours | 26.4 [23.5 to 32.6] | 28.2 [23.5 to 41.4]

3. Secondary Outcome: Post-discharge Nausea
Description: To be assessed based on patient diary completed daily for 1 week following discharge to home from the hospital
Time Frame: 1 week from discharge from hospital
Population: This analysis only possible with patients who successfully completed the post-discharge diary. Therefore, the participant number differs from the total patients enrolled.
Measure: Number; unit: percentage of subjects with PDN
Groups:
- Intervention Cohort: Patients undergoing maxillary surgery using the antiemetic anesthetic protocol who completed the post-discharge diary.
- Comparison Cohort: This arm was a retrospective comparison cohort treated at the same institution, managed per provider preference prior to protocol implementation, who completed the post-discharge diary
Arm/Group | Intervention Cohort | Comparison Cohort
Number analyzed (Participants) | 79 | 103
percentage of subjects with PDN | 72 | 60

4. Primary Outcome: Post-operative Vomiting
Time Frame: End of surgery to discharge from hospital
Measure: Number; unit: percentage of subjects with POV
Arm/Group | Intervention Cohort | Comparison Cohort
Number analyzed (Participants) | 93 | 137
percentage of subjects with POV | 11 | 28

5. Secondary Outcome: Post-discharge Vomiting
Time Frame: 1 week post discharge
Population: as for outcome 3
Measure: Number; unit: percentage of subjects with PDV
Arm/Group | Intervention Cohort | Comparison Cohort
Number analyzed (Participants) | 79 | 103
percentage of subjects with PDV | 22 | 29

ADVERSE EVENTS:
Groups:
- Intervention Cohort: Patients undergoing maxillary surgery using the antiemetic anesthesia protocol
Arm/Group | Intervention Cohort | Comparison Cohort
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/137
Other Adverse Events (participants affected / at risk) | 0/93 | 0/137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes